CLINICAL TRIAL: NCT05642975
Title: Comparing Ultrasound-Guided Suprainguinal Fascia Iliaca Block With Lumbar Erector Spinae Plane Block in Hip and Proximal Femur Fracture Surgery
Brief Title: Comparing Suprainguinal Fascia Iliaca Block With Erector Spinae Plane Block in Hip and Proximal Femur Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 11.2022.546
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Femur Fracture; Regional Anesthesia
Keywords: Postoperative Pain; Lumbar Erector Spinae Plane Block; Fascia Iliaca Block
MeSH Terms: conditions — Pain, Postoperative; Femoral Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suprainguinal Fascia Iliaca Block (Active Comparator): The probe was placed over the inguinal ligament in close proximity to the anterior superior iliac spine and oriented in the parasagittal plane. It was then moved inferomedially along the line of the inguinal ligament to visualize the 'bow-tie' sign. After confirming the needle's position, a total volume of 30 ml of bupivacaine 0.25% was injected.
  Spinal anesthesia was administered to the patients in a lateral position using 2.5 ml of 0.5% heavy bupivacaine at the L3-L4 level.
  Interventions: Procedure: Regional Block Comparison
- Erector Spinae Plane Block (Active Comparator): The L5, L4, and L3 transverse processes and erector spinae muscles posteriorly were identified using ultrasound. The curved 6-2 MHz transducer was initially placed at the mid-vertebral line in the sagittal plane and then shifted laterally to visualize the erector spinae muscle and transverse process of the L3 vertebra. A total volume of 40 ml of bupivacaine 0.25% was injected.
  Spinal anesthesia was administered to the patients in a lateral position using 2.5 ml of 0.5% heavy bupivacaine at the L3-L4 level.
  Interventions: Procedure: Regional Block Comparison
- Spinal Anesthesia Group (control) (Active Comparator): Spinal anesthesia was administered to the patients in a lateral position using 2.5 ml of 0.5% heavy bupivacaine at the L3-L4 level.
  Interventions: Procedure: Regional Block Comparison

INTERVENTIONS:
Procedure: Regional Block Comparison — Comparing postoperative pain and opioid consumption in groups

SUMMARY:
Most hip fractures occur in the elderly population. Opioid-related respiratory depression is more common in the elderly population but can cause severe brain damage or death. Reducing the amount of opioids administered before, during and after surgery by adding a regional block may increase the postoperative quality of recovery, reduce chronic pain syndromes, and may potentially facilitate the participation of patients in rehabilitation.

Despite their potential advantages, peripheral nerve blocks are still not widely used in people with hip fractures.

The primary objective of this study is to compare patients' postoperative pain scores and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, undergoing hip fracture surgery

Exclusion Criteria:

* Patients with solid organ dysfunction, chronic opioid or corticosteroid use, bleeding diathesis, patients receiving inpatient medication, patients with psychiatric disorders and patients who cannot be contacted after surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | 48 hours
  Comparing opioid consumption via Patient Controlled Analgesia (PCA) device

SECONDARY OUTCOMES:
Patient Satisfaction | 48 hours
  patient satisfaction score: 0: unsatisfied 5: fully satisfied
Complications Related to Pain Management | 48 hours
  complications such as hypothension, nausea, vomiting, itching
Postoperative Pain Scores | 48 hours
  Comparing pain scores with Numeric Rating Scale (NRS)
The lengths of ICU and hospital stays | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided